CLINICAL TRIAL: NCT01707680
Title: Non-interventional Comparison of Sedatives on Weaning From Mechanical Ventilation in Intensive Care Patients
Acronym: NICEWEAN
Status: Terminated | Type: Observational
Why Stopped: Halted due to slow recruitment
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 3005022; Dnr 2012/628-31/4 (Other: Ethical Review Board, Stockholm Region)
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Critical Illness
Keywords: weaning; mechanical ventilation; dexmedetomidine; propofol; midazolam
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dexmedetomidine: Here, patients to be included are those being sedated with dexmedetomidine as primary sedative.
  Interventions: Other: SOC
- Propofol: Here, patients to be included are those being sedated with propofol as primary sedative.
  Interventions: Other: SOC
- Midazolam: Here, patients to be included are those being sedated with midazolam as primary sedative
  Interventions: Other: SOC

INTERVENTIONS:
Other: SOC — Patient are given standard of care

SUMMARY:
The purpose of this study is to determine whether the use of different sedatives affect the weaning process from mechanical ventilation in intensive care patients.

DETAILED DESCRIPTION:
Traditionally patients with ongoing mechanical ventilation have been sedated to assure absence of pain, anxiety and to provide comfort. Unfortunately this approach might have negative consequences such as prolonged time for mechanical ventilation, length of stay in the ICU and hospital.

In this study, the investigators would like to investigate (in an exploratory way due to the non-interventional setup) whether weaning from mechanical ventilation will be affected by the choice of sedatives - including dexmedetomidine, midazolam and propofol. This study also aims at investigating how the choice of primary sedative will affect delirium/anxiety, need of other medications (sedatives, analgesics, anti-psychotics), quality of life after ICU and the presence of Post-Traumatic Stress Disorder. In addition, the investigators aim at receiving information from the caregivers on their ICU experience, as recent data imply that not only the ICU patient but also the caregiver suffer from PTSD after the ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to a general ICU ward
* ≥ 18years
* Intubated and mechanically ventilated for at least 24 hours
* Need of light to moderate sedation (corresponding to RASS 0 - (-3) or MAAS 2-3)
* Sedated with dexmedetomidine, midazolam and/or propofol
* Good knowledge in Swedish language
* Signed informed consent

Exclusion criteria:

* Lack of fulfilling prescribed sedation regime
* Estimated high risk of death during the study period, according to investigator (roughly equal to estimated mortality rate (EMR) > 80% )
* Tracheotomy
* Change in sedative drugs since the "fit for weaning" time point
* Use of other alpha-2 agonists (clonidine) during ICU stay
* Positive pregnancy test or currently lactating/ known pregnancy or lactation
* Participation in other study involving use of a pharmacologically active compound
* Patients with limitations in therapy
* Otherwise unable to fulfill the study, according to investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult general intensive care patients Need of mechanical ventilation >24 hours Need of light to moderate sedation
Sampling Method: Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2012-06-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
The time point from when the patient is considered "fit for weaning" to the actual time point for extubation | 30 days

SECONDARY OUTCOMES:
Time-point for patient being considered "fit for extubation" | 30 days
Total time in mechanical ventilation | 30 days
Extubation failure (re-intubation within 24 hours) | 24 hours
Anxiety/delirium assessments | 30 days
  RASS/MAAS sedation scales and ICDSC/CAM-ICU delirium assessments methods are used, as appropriate
Length of ICU stay (actual time of discharge) | 30 days
QoL (15D) | 2-4 months post-ICU discharge
Post-Traumatic Stress Disorder assessment - PTSS14 questionnaire | 2-4 months post-ICU discharge
  This assessment will be offered to the ICU patients but also to their caregivers.
Total duration of sedation | 30 days
Number of days using opioids | 30 days
Number of days using antipsychotic/neuroleptic drugs | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Carl-Johan Wickerts, MD, Principal Investigator — Danderyds Hospital, Danderyd, Sweden
Locations (3):
- Sweden (3):
  - Danderyds Hospital Anestesi- och intensivvårdskliniken, Danderyd
  - Örebro University Hospital, Anestesi- och intensivvårdskliniken, Örebro
  - Capio S:t Goran Hospital, Anestesikliniken, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nunes SL, Forsberg S, Blomqvist H, Berggren L, Sorberg M, Sarapohja T, Wickerts CJ. Effect of Sedation Regimen on Weaning from Mechanical Ventilation in the Intensive Care Unit. Clin Drug Investig. 2018 Jun;38(6):535-543. doi: 10.1007/s40261-018-0636-2. PMID 29502195